CLINICAL TRIAL: NCT03811977
Title: The Effect of 12-Week Dietary Intake of Lutein on Minimal Erythema Dose and Other Skin Parameters: Randomised Double-Blind Placebo Controlled Study
Brief Title: The Effect of 12-Week Dietary Intake of Lutein on Minimal Erythema Dose and Other Skin Parameters
Acronym: VIST Lutein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: European Regional Development Fund (Other); Ministry of Education, Science and Sport, Republic of Slovenia (Unknown); Dermatologija Bartenjev Rogl (Unknown); Slovenian Research Agency (Other); Valens Int. d.o.o., Slovenija (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIST F4F Lutein-MED 01-2018
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-01

CONDITIONS: Minimal Erythema Dose; Skin Viscoelasticity; Dermis Density

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Test group will receive investigational product - lutein syrup (2 mg/mL; daily dose 20 mg). Participants in this group will test continuous administration of investigational product for 12 weeks.
  Interventions: Dietary Supplement: Lutein syrup
- Placebo group (Placebo Comparator): Placebo group will receive placebo product - placebo syrup (lutein 0 mg/mL; daily dose 0 mg). Continuous administration of placebo product for 12 weeks.
  Interventions: Dietary Supplement: Placebo syrup

INTERVENTIONS:
Dietary Supplement: Lutein syrup — 12- week dietary supplementation with lutein syrup (20 mg lutein/day)
  Arms: Test group
Dietary Supplement: Placebo syrup — 12- week dietary supplementation with placebo syrup (0 mg lutein/day)
  Arms: Placebo group

SUMMARY:
The double-center, randomized, placebo-controlled, one-period effectiveness study will include 30 subjects (women, aged between 25 to 55 years, Fitzpatrick phototype II and III). Subjects will be divided in two groups, 15 in each. One group (test group) will receive investigational product - lutein syrup (4 mg/mL; daily dose 20 mg) and the other (placebo group) placebo syrup. Participants will test continuous administration of placebo or investigational product for 12 weeks in order to demonstrate and assess multiple-dose effects. The primary objective is to assess the photoprotective potential of the investigational product in relation to placebo product. The secondary objectives are to assess effects of investigational product on dermis density and skin viscoelasticity after 12 weeks of dietary supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian female volunteers aged between 25 and 55 years at the time of the signature of Informed consent form (ICF),
* Signed Informed consent form (ICF),
* Fitzpatrick skin phototypes II and III,
* No skin pigmentation disorders,
* In good health condition,
* Willingness to avoid a consumption of any food supplements containing carotenes or other antioxidants during the study,
* Willingness to avoid the sun, tanning beds and tanning products on the gluteal area during the study,
* Willingness to follow all study procedures and keeping a diary for during the study (to follow their compliance and palatability),
* No changes in dietary habits or dietary supplements in last month prior to inclusion.
* No changes in cosmetic facial and body care routine in last month prior to inclusion on measurement areas.

Exclusion Criteria:

* Pregnancy or breastfeeding,
* Known or suspected allergy to any ingredient of the tested products or UV radiation,
* Changes in dietary habits and dietary supplementation in last month prior to inclusion,
* Veganism,
* Changes in cosmetic facial and body care routine in last month prior to inclusion.
* Diagnosed and uncontrolled/untreated/unregulated disease,
* Any clinically significant history of serious metabolic disease, digestive tract disease, liver disease, kidney disease, haematological disease.
* Acute skin diseases,
* Regular consumption of food supplements containing carotenoids or other antioxidants in last month before inclusion into the study.
* Invasive rejuvenation treatments (e.g. needle rollers, needle mesotherapy, deep/medium-deep chemical peels etc.) in last 6 months prior to study entry,
* Non-invasive rejuvenation treatments (e.g. radiofrequency, electrotherapy, ultrasound therapy) in last 2 months prior to study entry,
* Gluteal hyperpigmentation,
* Mental incapacity that precludes adequate understanding or cooperation

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Photoprotective potential of the investigational product in relation to placebo product assessed through measurements of minimal erythema dose | 12 weeks
  The primary objective is to assess the photoprotective potential of the investigational product in relation to placebo product. It will be assessed through measurements of minimal erythema dose with MED Tester using UVB irradiation. Significant change of minimal erythema dose from baseline in test group, in comparison to placebo group, after 12 weeks of dietary supplementation with study product is expected.

SECONDARY OUTCOMES:
Influence of investigational product in relation to placebo product on dermis density assessed through dermis intensity measurement | 12 weeks
  Significant change of dermis density from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected. Dermis density will be assessed through ultrasonographic dermis intensity measurement.
Influence of the investigational product in relation to placebo product on skin elasticity assessed through measurements of viscoelasticity | 12 weeks
  For assessments of skin elasticity viscoelasticity measurements will be performed. Significant change of skin easticity from baseline in test group, in comparison to placebo group after 12 weeks of dietary supplementation with study product is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, Study Director — Head of Research Group
Locations (1):
- Higher School of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No